CLINICAL TRIAL: NCT05286749
Title: Community Health Outreach to Increase Cervical Cancer Education and Self-Collection Screening (CHOICESS) Program for Southeast Asian Immigrant and Refugee Women in Wisconsin
Brief Title: Cervical Cancer Self-Collection for Southeast Asian Immigrant and Refugee Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Milwaukee Consortium for Hmong Health (MCHH) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2021-1525; Protocol Version 8/8/2023 (Other: UW Madison); UW21142 (Other: UWCCC); A532050 (Other: UW Madison)
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Cervical Cancer Screening
Keywords: self-collection; community health workers

STUDY DESIGN:
Intervention Model Description: Workshops are randomized to either a control or intervention group
Who Masked: Participant
Masking Description: Participants will be informed of random assignment into two groups. Participants will not be aware of which group they belong to. Participants in the control group are initially only provided educational materials about the standard of care for cervical cancer screening and offered clinician-collection for screening as the recommended method. Whereas the intervention group is provided additional materials about self-collection in the core educational material and is offered the Evalyn Device for self-collection as a screening option immediately at the end of the workshop. All participants will be made aware during a debrief session at the end of the study about what information could not be given at the time of consenting, and why they could not be told at that time.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Control (Active Comparator): Participants take a workshop where they are provided education on standard-of-care for cervical cancer screening such as pap smear and HPV testing through clinician-collection methods using speculum and cervical swabs.
  Interventions: Procedure: Workshop plus Clinician-Collected Cervical Swab
- Intervention (Experimental): Participants take a workshop where they are provided all the same education as control as well as additional education on self-collection for HPV-only testing using vaginal swab as an additional method.
  Interventions: Device: Workshop plus Participant-Collected Cervical Swab; Diagnostic Test: HPV testing on Participant-Collected Cervical Swab Samples

INTERVENTIONS:
Procedure: Workshop plus Clinician-Collected Cervical Swab — clinician-collection methods using speculum and cervical swabs
  Arms: Control
Device: Workshop plus Participant-Collected Cervical Swab — Evalyn® Brush (Rovers® Medical Devices, Netherlands)
  Arms: Intervention
Diagnostic Test: HPV testing on Participant-Collected Cervical Swab Samples — Roche Cobas4800 HPV Test System (Roche Molecular Systems Inc., Rotkreuz, Switzerland)
  Arms: Intervention

SUMMARY:
The primary purpose of this study is to determine whether educational workshops paired with self-collected high-risk human papillomaviruses (hrHPV) screening will increase participation in cervical cancer screening among Southeast Asian Immigrant and Refugee populations in Wisconsin compared with offering clinician collected screening (total sample size: 250 participants). The investigators hypothesize that participation in cervical cancer screening will be higher among women in the intervention group as compared to the control group.

DETAILED DESCRIPTION:
The effectiveness of offering self-collection sampling options to Southeast Asian refugee and immigrant populations to improve cervical cancer screening participation has not been investigated. The Milwaukee Consortium for Hmong Health (MCHH), supported by the Well Woman Program, has had success increasing participation in breast cancer screening through outreach and education activities. However, it continues to have limited success engaging women in cervical cancer screening. The investigators have established a partnership with MCHH to develop innovative cervical cancer workshops that combine community health worker (CHW)-led engagement with self-collected hrHPV screening, with the primary objective of increasing participation, awareness, and engagement in cervical cancer screening and treatment activities among this population.

Research Intervention: Control workshops are workshops where participants are provided education on standard-of-care for cervical cancer screening such as pap smear and HPV testing through clinician-collection methods using speculum and cervical swabs. Intervention workshops are workshops where participants are provided all the same education as control as well as additional education on self-collection for HPV-only testing using vaginal swab as an additional method. After each workshop, each group will be offered to participate in their assigned group's screening method (clinician-collected or self-collected).

* Primary Objective: To evaluate whether educational workshops paired with self-collected hrHPV screening will increase participation in cervical cancer screening among Southeast Asian refugee and immigrant populations in Wisconsin compared with offering clinician-collected screening.
* Secondary Objectives: To evaluate participant satisfaction with the educational workshops using satisfaction surveys.

ELIGIBILITY:
Inclusion Criteria:

* Fluent understanding in English, Hmong, Karen, Burmese, or Karenni

Exclusion Criteria:

* Prior hysterectomy
* Impaired decision-making capacity
* Pregnancy

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2022-08-13 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Dalby, MD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- MCHH's Community Center, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Intervention
Started | 75 | 78
Completed | 75 | 78
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 75 | 78 | 153
Age, Customized [Count of Participants; unit: Participants]
  25 to 35 years | 26 | 20 | 46
  36 to 45 years | 19 | 23 | 42
  46 to 55 years | 15 | 19 | 34
  56 to 65 years | 15 | 16 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 78 | 153
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic Group: Burmese | 18 | 19 | 37
  Ethnic Group: Hmong | 17 | 18 | 35
  Ethnic Group: Karenn | 13 | 15 | 28
  Ethnic Group: Karenni | 27 | 26 | 53
Region of Enrollment [Number; unit: participants]
  United States | 75 | 78 | 153
Highest Level of Education [Count of Participants; unit: Participants]
  College or Above | 10 | 8 | 18
  High School or Less | 27 | 34 | 61
  None | 8 | 13 | 21
  No Answer | 30 | 23 | 53
Employment Status [Count of Participants; unit: Participants]
  Employed | 34 | 36 | 70
  Unemployed | 30 | 30 | 60
  No Answer | 11 | 12 | 23
Marital Status [Count of Participants; unit: Participants]
  Married | 50 | 48 | 98
  Single | 20 | 16 | 36
  No Answer | 5 | 14 | 19
Insurance Status [Count of Participants; unit: Participants]
  Medicaid | 48 | 42 | 90
  Medicare | 0 | 3 | 3
  Private Insurance | 18 | 19 | 37
  No insurance | 9 | 10 | 19
  No answer | 0 | 4 | 4
Birth Country [Count of Participants; unit: Participants]
  United States | 5 | 1 | 6
  Outside of the United States | 70 | 77 | 147
Years Living in the US [Count of Participants; unit: Participants]
  5 years or less | 8 | 4 | 12
  6 to 10 years | 15 | 21 | 36
  11 to 30 years | 24 | 34 | 58
  more than 30 years | 15 | 10 | 25
  No Answer | 13 | 9 | 22
Comfort with Written English [Count of Participants; unit: Participants]
  Very comfortable | 10 | 5 | 15
  Somewhat comfortable | 6 | 6 | 12
  Neutral | 19 | 19 | 38
  Somewhat uncomfortable | 11 | 14 | 25
  Not at all comfortable | 27 | 32 | 59
  No Answer | 2 | 2 | 4
Comfort with Oral (heard) English [Count of Participants; unit: Participants]
  Very comfortable | 9 | 7 | 16
  Somewhat comfortable | 9 | 6 | 15
  Neutral | 17 | 16 | 33
  Somewhat uncomfortable | 13 | 20 | 33
  Not at all comfortable | 25 | 26 | 51
  No Answer | 2 | 3 | 5
Comfort with Written Native Language [Count of Participants; unit: Participants]
  Very comfortable | 24 | 29 | 53
  Somewhat comfortable | 12 | 9 | 21
  Neutral | 9 | 11 | 20
  Somewhat uncomfortable | 5 | 6 | 11
  Not at all comfortable | 22 | 19 | 41
  No answer | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Obtain or Self-Report Future Desire for Cervical Cancer Screening
Description: The results will be reported through summary statistics of the number of participants in each group subsequently engaging or seeking out cervical cancer screening either through services offered after workshop education or self-reported desire to follow up through their community health care provider.
Time Frame: up to 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 75 | 78
Participants | 59 | 71

2. Secondary Outcome: Participant Satisfaction With Educational Workshops Survey Scores
Description: Participant satisfaction with the educational workshops will be assessed using mixed methods satisfaction surveys. 4-items on the pre- and post-workshop surveys scored on a 5 point likert scale from 1 (not likely) to 5 (very likely) for a total possible range of scores from 1 to 5 where higher scores are a proxy for positive workshop impact on participant. Additional items will include open ended questions on satisfaction.
Time Frame: up to 1 day (pre workshop and post-workshop, up to 3 hours between surveys)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 75 | 78
score on a scale
  Likelihood to get pap in future | 4.6 (0.854) | 4.44 (1.112)
  Likelihood to spread word about screenings to family/friends | 4.76 (0.654) | 4.63 (0.913)
  Likelihood to encourage your family members to get screened | 4.71 (0.653) | 4.74 (0.653)
  Practice healthy behaviors to reduce risk | 4.73 (0.664) | 4.88 (0.394)

3. Secondary Outcome: Number of Participants Willing to Use HPV Self-collect Device for Their Cervical Cancer Screening
Description: General willingness to use a HPV self-collect device at home and/or as the preferred collection method for cervical cancer screening, assessed via mixed methods survey.
Time Frame: up to 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 75 | 78
Participants | 6 | 1

ADVERSE EVENTS:
Time Frame: data collected during 1 study visit, up to 3 hours
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/78
Other Adverse Events (participants affected / at risk) | 0/75 | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT05286749/Prot_SAP_000.pdf